CLINICAL TRIAL: NCT03785327
Title: Improving Social Interaction for Adolescents With Autism During the Transition to Adulthood
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID disrupted data collection
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Noah Sasson, Associate Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1806799
Record Dates: First submitted 2018-10-29; First posted 2018-12-24 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Autism Spectrum Disorder; Typical Development
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Autistic participants were going to be recruited for an active or sham tDCS session. However, no participants were enrolled in these conditions due to COVID.
  TD participants were assigned to receive or not receive a training session.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Active anodal tDCS (Experimental): Active anodal tDCS followed by behavioral testing Intervention: Device: active anodal tDCS
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): Sham tDCS followed by behavioral testing Intervention: Device: sham tDCS
  Interventions: Device: tDCS
- Autism Training Program (Experimental): Training program designed to increase autism understanding followed by behavioral testing Intervention:Training program
  Interventions: Behavioral: Autism Training
- Social interaction without intervention (No Intervention): Control condition: Behavioral testing without an intervention component

INTERVENTIONS:
Device: tDCS — Participants either complete active and sham tDCS sessions one week apart or an autism training program.
  Arms: Active anodal tDCS; Sham tDCS
Behavioral: Autism Training — Autism Information Presentation developed by Dr. Grace Iarocci's Autism & Developmental Disorders Lab at Simon Fraser University
  Arms: Autism Training Program

SUMMARY:
This study compares the efficacy of two intervention strategies for improving social outcomes for autistic adolescents and young adults when interacting with unfamiliar non-autistic peers.

DETAILED DESCRIPTION:
Intellectually-capable older adolescents and young adults with autism spectrum disorder (ASD) often struggle to secure and maintain employment, succeed in college, or develop satisfying personal and professional relationships. Current psychosocial interventions for this population have produced limited effects on real-world functioning. These programs typically seek to improve social skill and understanding with the hope that these abilities will translate to better functioning and are often effective at increasing knowledge of social rules and norms,yet these improvements frequently do not translate to better social and life outcomes in the real world. One reason for their limited efficacy may be that the mechanisms involved in real-life social interaction continue to be poorly understood for this population. The current study is designed to specify the factors that predict more or less favorable social outcomes for autistic adolescents and young adults when interacting with an unfamiliar, non-autistic peer, and test a multifaceted intervention for improving these outcomes. The intervention will target both brain and behavior, not only in the individual with ASD but also in their typically-developing (TD) partners. For TD participants, the efficacy of a training program will be tested to determine if social experiences for older adolescents with ASD can be improved by increasing knowledge, acceptance, and understanding of autism among TD individuals. For the participants with ASD, this study will test the efficacy of an innovative, non-invasive neurostimulation session using Transcranial Direct Current Stimulation (tDCS) to target social brain regions involved in perspective-taking and social reciprocity. Social outcomes for each intervention will be compared to a "no intervention" control condition, and to each other, to provide a comprehensive examination of intrinsic and extrinsic factors contributing to social interaction quality for autistic adolescents and young adults.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-21
* DSM-IV-TR or DSM-5 diagnosis of an Autism Spectrum Disorder
* IQ>70

Exclusion Criteria:

* Presence or history intellectual impairment (defined as IQ <70)
* Presence or history of medical, cardiac, or neurological disorders that may affect brain function (e.g., cardiac disease, endocrine disorders, renal disease, pulmonary disease, history of seizures or head trauma with unconsciousness for a period of 15 minutes or greater or CNS tumors)
* Presence of sensory limitation including visual (e.g., blindness, glaucoma, vision uncorrectable to 20/40) or hearing (e.g. hearing loss) impairments that interfere with assessment
* Not proficient in English
* Presence of substance abuse in the past one month
* Presence of substance dependence not in remission for the past six months
* Contraindications for tDCS (e.g., pregnancy or implanted devices such as pace maker)

Ages: 18 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-09-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Dallas, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Anodal tDCS | Sham tDCS | Autism Training Program | Social Interaction Without Intervention
Started | 0 | 0 | 38 | 40
Completed | 0 | 0 | 38 | 40
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Active and Sham tDCS were terminated before beginning due to COVID
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Anodal tDCS | Sham tDCS | Autism Training Program | Social Interaction Without Intervention | Total
Number analyzed (Participants) | 0 | 0 | 38 | 40 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] |  |  | 20.26 (1.79) | 20.63 (1.75) | 20.45 (1.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  | 0 | 0 | 0
  Male |  |  | 38 | 40 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  |  | 2 | 8 | 10
  Not Hispanic or Latino |  |  | 36 | 32 | 68
  Unknown or Not Reported |  |  | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  |  | 38 | 40 | 78

OUTCOME MEASURES:

1. Primary Outcome: Subjective Social Interaction Quality
Description: Non-autistic participants social interest in autistic partners as measured by the First Impression Scale (Sasson et al., 2017). Four items, each scored on a Likert Scale from 1 to 4 in which higher values indicate greater social interest, are averaged to produce a social interest composite that serves as the primary outcome measure of the non-autistic participant's social interest in their autistic conversation partner.
Time Frame: Interaction with unfamiliar partner occurs immediately following the autism training; self-report measure given immediately after the interaction, duration of completion averages around 2 minutes
Population: Zero participants are listed for the Active and Sham tDCS arms because these arms were terminated before data collection began.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Anodal tDCS | Sham tDCS | Autism Training Program | Social Interaction Without Intervention
Number analyzed (Participants) | 0 | 0 | 38 | 40
units on a scale |  |  | 2.74 (0.45) | 2.45 (0.61)

ADVERSE EVENTS:
Time Frame: 1-2 hours, which is the average duration of participation for each individual participant in the "Autism Training Program" arm and "Social Interaction without Intervention " arm; participants were not enrolled in the "active and sham tCDS" arms.
Description: Zero participants are listed as at risk in the active and sham tCDS arms because these arms were terminated before beginning. No participants were tested in them.
Arm/Group | Active Anodal tDCS | Sham tDCS | Autism Training Program | Social Interaction Without Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/38 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/38 | 0/40
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/38 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT03785327/Prot_SAP_000.pdf